CLINICAL TRIAL: NCT06860386
Title: A Phase II Study Assessing the Feasibility and Clinical Efficacy of Adaptive Immunotherapy Combination With VEGFR-TKI in Patients With Advanced Renal Cell Carcinoma
Brief Title: Study of Adaptive Immunotherapy With VEGFR-TKI in Patients With Advanced RCC
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: Funding unavailable
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-23473
Record Dates: First submitted 2025-03-04; First posted 2025-03-06 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Renal Cell Carcinoma; Clear Cell Renal Cell Carcinoma
Keywords: Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — pembrolizumab; Axitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Adaptive Dosing pembro-axi (Experimental): In therapy naïve mccRCC patients, a standard dose of pembrolizumb will be given at 200 mg iv every 3 weeks, with axitinib given orally 5 mg twice daily.
  After 9 weeks, subjects will undergo the first response assessment as well as the therapy portion of the trial if they have 20% response per RECIST criteria.
  During adaptive dosing with pembro-axi, imaging is conducted every 9 weeks. Treatment is held until the tumor has returned to its baseline size or greater per RECIST 1.1, then restarted until a tumor reduction of at least 20% occurs.
  Therapy cycles on and off in this manner continue as the tumor shrinks and grows until confirmed progression of disease while on therapy.
  Interventions: Drug: Pembrolizumab; Drug: Axitinib

INTERVENTIONS:
Drug: Pembrolizumab — 200 mg every 3 weeks IV infusion (Q3W + or -3 days)
  Other Names: KEYTRUDA
Drug: Axitinib — 5 mg twice daily (BID) by mouth
  Other Names: INLYTA

SUMMARY:
This is a Phase II Clinical Trial that will evaluate the use of adaptive dosing of pembro-axi in patients with Metastatic Clear Cell Renal Cell Carcinoma (mccRCC).

ELIGIBILITY:
Inclusion Criteria:

* Unresectable advanced or metastatic Renal Cell Carcinoma (RCC) to include only predominant clear cell histology.
* Age ≥ 18 years or older at time of signing informed consent.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of ≤ 2 within 28 days prior to registration.
* Availability of formalin-fixed, paraffin-embedded (FFPE) archival tumor specimens, when available, and willingness of the subject to undergo fresh tumor biopsy prior to treatment initiation if archival tissue not available.

  * If a target lesion is biopsied at screening, this lesion must be followed as non-target lesion after the biopsy unless it is the patient's only target lesion.
  * If there is only one target lesion, it should be followed as a target lesion regardless.
  * The archival specimen must contain adequate viable tumor tissue.
  * The specimen may consist of a tissue block (preferred and should contain the highest grade of tumor) or at least 30 unstained serial sections. Fine needle aspiration/ biopsy, brushings, cell pellet from pleural effusion, bone lesion, bone marrow aspirate/biopsy are not acceptable.
* Have had no prior systemic therapy (treatment naïve) for Metastatic Clear Cell Renal Cell Carcinoma (mccRCC). Prior neoadjuvant or adjuvant therapy received for localized ccRCC is not allowed.
* Measurable disease as defined by Response Evaluation Criteria In Solid Tumors RECIST 1.1 within 28 days prior to registration.
* Must demonstrate adequate hematological, hepatic and kidney organ function with all screening labs to be obtained within 28 days prior to first study treatment.
* Females of childbearing potential must have a negative serum pregnancy test within 28 days prior to registration. NOTE: Females are considered of childbearing potential unless they are surgically sterile (have undergone a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or they are naturally postmenopausal for at least 12 consecutive months.
* Females of childbearing potential and males must be willing to abstain from heterosexual activity or to use 2 forms of effective methods of contraception from the time of informed consent until 150 days after treatment discontinuation for females and 210 days after treatment discontinuation for males. The two contraception methods can be comprised of two barrier methods, or a barrier method plus a hormonal method.
* As determined by the enrolling physician or protocol designee, must have ability to comprehend and the willingness to sign written informed consent, and comply with study procedures for entire length of study to be eligible for study participation.
* Patients with well-controlled Hepatitis B, Hepatitis C, or HIV will be considered eligible.

Exclusion Criteria:

* Has had major surgery within 4 weeks and/or has received radiation therapy within 2 weeks prior to Cycle 1, Day 1 (C1D1).
* Has received prior systemic anti-cancer therapy for RCC (e.g., VEGF/VEGFR, chemotherapy or mTOR-targeting agents). Note: Prior neoadjuvant/adjuvant therapy for ccRCC is acceptable if last dose was received more than 3 months from start of C1 D1.
* Has a history of severe hypersensitivity reaction (e.g., generalized rash/erythema hypotension, bronchospasm, angioedema, or anaphylaxis) to axitinib or pembrolizumab.
* Has a diagnosis of immunodeficiency OR is receiving a systemic steroid therapy exceeding physiologic corticosteroid dose or any other form of immunosuppressive therapy within 7 days prior to C1D1.

Note: Subjects with vitiligo, Sjögren's syndrome, Type 1 diabetes, or resolved childhood asthma/atopy will not be excluded from the study. Subjects requiring intermittent use of bronchodilators, inhaled steroids, or local steroid injections will not be excluded from the study. Subjects with hypothyroidism, or adrenal or pituitary insufficiency who are stable on hormone replacement will not be excluded from the study.

* Has a known additional malignancy that has progressed or has required active treatment in the last 1 year. Note: Basal cell carcinoma of the skin, squamous cell carcinoma of the skin, superficial bladder cancer, or carcinoma in situ such as breast cancer in situ are acceptable if they have undergone potentially curative therapy.
* Has known active CNS metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are radiologically stable, i.e., without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to C1D1.
* Has a history of (non-infectious) pneumonitis that required steroids in the past 6 months or current pneumonitis.
* Has an active infection requiring systemic therapy.
* Has a known history of Human Immunodeficiency Virus (HIV) infection (e.g. HIV 1 and/or 2 antibodies), that is not well controlled.
* Has a known history of Hepatitis B (e.g., Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (e.g., HCV RNA [qualitative] is detected), that is not well controlled.
* Has a clinically significant gastrointestinal (GI) abnormality including: Malabsorption, total gastric resection, or any other condition that might affect the absorption of orally taken medication. Active GI bleeding, as evidenced by hematemesis, hematochezia or melena in the past 3 months without evidence of resolution documented by endoscopy or colonoscopy. Intraluminal metastatic lesion with suspected bleeding, inflammatory bowel disease, ulcerative colitis or other GI condition associated with increased risk of perforation.
* 12-lead ECG will be performed during screening. If the initial QTcF is found to be > 500 msec, two additional EKGs separated by at least 3 minutes should be performed. If the average of these three consecutive results for QTcF is ≤ 500 msec, the subject meets eligibility in this regard.
* Has a known history of any of the following cardiovascular conditions within 6 months of C1D1 of therapy:

  * Myocardial infarction
  * Unstable angina pectoris
  * Cardiac angioplasty or stenting
  * Coronary/peripheral artery bypass graft
  * Class III or IV congestive heart failure per New York Heart Association
  * Cerebrovascular accident or transient ischemic attack
* Has poorly controlled hypertension defined as systolic blood pressure (SBP) ≥ 160 mmHg and/or diastolic blood pressure (DBP) ≥ 90 mmHg. Subjects with initial screening BP ≥160/90 mmHg can be treated with anti-hypertensive medication to achieve a well-controlled status and are eligible with reassessed SBP/DBP of < 150/95 mm Hg.
* Has evidence of inadequate wound healing or active bleeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-02-25 (Actual); Primary Completion 2028-02 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Recruitment Rate Feasibility | Up to 36 Months
  Measured as the percentage of eligible patients with a >20% tumor response who consent to participate in the adaptive therapy.
  Successful enrollment if at least 70% of eligible patients agree to participate in the adaptive therapy
Progression Free Survival (PFS) | Up to 12 Months
  Measured from the start of treatment until the point of disease progression or death from any cause.

SECONDARY OUTCOMES:
Persistent Disease Control | Up to 36 Months
  Measured as the proportion of patients who complete adaptive therapy and do not requiring disease re-initiation for more than 12 months after therapy discontinuation.
Overall Survival (OS) | Up to 36 Months
  Measured as time from date of enrollment to death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Jon Chatzkel, MD, Principal Investigator — Moffitt Cancer Center
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States

REFERENCES:
- See also: Moffitt Cancer Center Clinical Trials Website — http://www.moffitt.org/clinical-trials-research/clinical-trials/